CLINICAL TRIAL: NCT01355874
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Treatment Group, Multicenter Efficacy and Safety Study of Intra-Anal Application of Iferanserin (10 mg) as a 0.5% Ointment in Subjects With Symptomatic Internal Hemorrhoids
Brief Title: Efficacy and Safety Study to Treat Subjects With Symptomatic Internal Hemorrhoids
Acronym: VEN309
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The primary endpoint was not met on the double blind data
Sponsor: Ventrus Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VEN 309-Hem-SE3-001
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2012-07

CONDITIONS: Internal Hemorrhoids
Keywords: Internal Symptomatic Hemorrhoids
MeSH Terms: interventions — iferanserin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Iferanserin (Experimental)
  Interventions: Drug: Iferanserin
- Placebo (Experimental)
  Interventions: Drug: Placebo
- Iferanserin + Placebo (Experimental)
  Interventions: Drug: Iferanserin + Placebo

INTERVENTIONS:
Drug: Iferanserin — 0.5% iferanserin ointment (containing 10 mg of iferanserin) BID for 14 days during double blind.
  Arms: Iferanserin
Drug: Placebo — Placebo ointment BID for 14 days during double blind.
  Arms: Placebo
Drug: Iferanserin + Placebo — 0.5% iferanserin ointment (containing 10 mg of iferanserin) BID for 7 days followed by placebo ointment BID for 7 days during the double blind.
  Arms: Iferanserin + Placebo

SUMMARY:
Primary Objective:

To evaluate the effect of iferanserin ointment on cessation of bleeding when administered intra-anally twice daily (BID) for 7 or 14 days in subjects with symptomatic internal hemorrhoids.

Methodology:

Double-Blind: Phase 3, multicenter, double-blind, randomized, parallel group, placebo-controlled part of the study. Extension: Multicenter, open-label part of the study.

Study Treatment Duration:

Double-Blind: 28 days (14-day treatment period and a 14-day follow-up period). Extension: 12 months (open-label part of the study in which there will be a scheduled visit every three months. Subjects who have recurrence(s) of their symptomatic internal hemorrhoids will be treated with open-label iferanserin for 7 days followed by a 21-day follow-up period).

Criteria for Evaluation:

Primary Endpoint:

The primary endpoint is the cessation of bleeding by the end of Day 7 that persists for the remainder of the treatment period (through Day 14).

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the effect of iferanserin ointment on cessation of bleeding when administered intra-anally twice daily (BID) for 7 or 14 days in subjects with symptomatic internal hemorrhoids. Safety Secondary Objective To determine the safety of iferanserin ointment administered intra-anally BID for 7 or 14 days in subjects with symptomatic internal hemorrhoids.

Exploratory Objectives:

To evaluate the frequency of recurrence of bleeding in subjects with symptomatic internal hemorrhoids. To evaluate time to bleeding recurrence in subjects with symptomatic internal hemorrhoids. To evaluate efficacy of iferanserin ointment in the treatment of recurrence when administered intra-anally BID for 7 days in subjects with symptomatic internal hemorrhoids. To evaluate the parameters of the Symptom Satisfaction Questionnaire

Methodology:

Double-Blind: Phase 3, multicenter, double-blind, randomized, parallel group, placebo-controlled part of the study. Extension: Multicenter, open-label part of the study.

Criteria for Evaluation:

Primary Endpoint:

The primary endpoint is the cessation of bleeding by the end of Day 7 that persists for the remainder of the treatment period (through Day 14).

Secondary Endpoints:

Key Secondary Endpoints Cessation of itching by the end of Day 7 that persists for the remainder of the treatment period (through Day 14). Cessation of pain by the end of Day 7 that persists for the remainder of the treatment period (through Day 14). Safety Secondary Endpoints Adverse events (AEs). Serious Adverse events (SAEs). Physical examination. Hematology, serum chemistry, and urinalysis. Vital signs. Electrocardiogram.

Exploratory Endpoints:

Bleeding recurrence rate of symptomatic internal hemorrhoids. Time to bleeding recurrence of symptomatic internal hemorrhoids. Response to open-label iferanserin ointment in the treatment of recurrence of symptomatic internal hemorrhoids. Overall improvement score for the parameters of the Symptom Satisfaction Questionnaire.

ELIGIBILITY:
1.1 Inclusion Criteria for Double-Blind and Recurrence

1. Males or non-pregnant females, aged ≥ 18 to ≤ 75 years.
2. Symptomatic internal hemorrhoids, Grades I-III by direct anoscopic visualization (anoscopic visualization not required if Grade determined by colonoscopy within 28 days prior to Day 1).
3. Bleeding from hemorrhoids for two consecutive days prior to randomization (Day 1).

   • For females experiencing menses, on the two days prior to randomization they must confirm that blood is from the anus and not from their menses by gently inserting a cotton swab into the anus after attempting a bowel movement; and they must see blood on the cotton swab for the two consecutive days prior to randomization to meet the inclusion criteria.
4. Itching OR pain for two consecutive days prior to randomization (Day 1).
5. Able to attempt bowel movements daily (defined as trying to have a bowel movement while sitting on the toilet for at least a few minutes, at least once daily, whether or not you feel the need to have a bowel movement that day).
6. Body mass index of ≥ 18.5 to ≤ 36 kg/m2.
7. Female of non-childbearing potential, including any female who: a) has had a hysterectomy, b) has had a bilateral oophorectomy, c) has had a bilateral tubal ligation or d) is post menopausal (demonstration of total cessation of menses for ≥ 1 year from the date of the screening visit).
8. Females of child bearing potential who agree to use two forms of contraception, one of which must be a barrier method, during the full duration of the study.
9. Able to communicate adequately with the investigator and to comply with the requirements for the entire study.
10. Capable of using the IVRS and adequately communicate comprehension of IVRS questions to the investigator.
11. Capable of and freely willing to provide written informed consent prior to participating in the study.

1. 1.2 Exclusion Criteria for Double-Blind and Recurrence

1. Grade IV internal hemorrhoids.
2. Age ≥ 40 years, with no complete colon evaluation within three years.
3. Age < 40 years, with no sigmoidoscopy or complete colon evaluation within three years.
4. Age < 40 years, with any of the following and no complete colon evaluation within two years; or age ≥ 40 years, with any of the following and no complete colon evaluation within one year:

   * History of adenomatous polyps.
   * Family history of either colorectal cancer or colorectal adenomas diagnosed in a first-degree relative before age 60.
   * Family history or genetic testing indicating the presence of one of two hereditary syndromes.
5. Malignancy within 5 years prior to Day 1(with the exception of treated basal cell/squamous cell carcinoma of the skin).
6. History of inflammatory bowel disease.
7. History of irritable bowel syndrome with constipation or diarrhea.
8. Previous surgical or instrumental treatment of internal hemorrhoids.
9. Clinical evidence or history of fecal incontinence.
10. Current thrombosed internal or external hemorrhoid(s).
11. Clinical evidence or history of anal fissure.
12. Clinical evidence or history of anal fistula.
13. AST/ALT > 3x ULN.
14. Hemoglobin < 10.0 g/dL.
15. Selective serotonin reuptake inhibitors within 28 days prior to Day 1.
16. Tamoxifen within 28 days prior to Day 1.
17. Laxatives (unless maintained on a stable dose of the medication for ≥ 60 days prior to Day 1).
18. Anticoagulants (e.g., coumadin, heparinoids, dabigatran) within 90 days prior to Day 1.
19. Anti-platelet agents or low dose aspirin (unless maintained on the medication for ≥ 90 days prior to Day 1).
20. Over the counter or prescription anti-hemorrhoid agents (including herbal supplements) within 14 days prior to Day 1.
21. Topical anesthetics within 14 days prior to Day 1.
22. Chronic use of analgesics (e.g., opioids, acetaminophen, aspirin, NSAIDS, cox-2 inhibitors, etc).
23. Any investigational agents within 28 days prior to Day 1 (with the exception of iferanserin for recurrence).
24. Anti-TNF agents within 6 months prior to Day 1.
25. Oral or parenteral steroids within 28 days prior to Day 1.
26. Use of anal, intra-anal, or intra-rectal steroids within 28 days prior to Day 1.
27. Expected to have a planned interventional and/or surgical procedure that requires hospitalization, colonoscopy, or sigmoidoscopy (colonoscopy or sigmoidoscopy during the screening period is acceptable).
28. Following concomitant disease state:

    * Clinical evidence or history of significant cardiovascular disease including arrhythmias, clinically significant ECG abnormalities, myocardial infarction, stroke, congestive heart failure (greater than class II), and valve disease or abnormalities.
    * Asthma currently requiring treatment (with the exception of infrequent use of rescue inhaler).
    * Clinical evidence or history of chronic renal failure (greater than Stage III).
    * Clinical evidence or history of gastric ulcer, duodenal ulcer, or pancreatitis.
    * Clinical evidence or history of hematological disease.
    * Clinical evidence or history of neurological disease.
    * Acute infection currently requiring treatment.
    * Clinical evidence or history of chronic infectious disease.
29. Major organ transplant.
30. Any disease or prior surgery that may interfere with the subject successfully completing the study.
31. History of any prior anal or rectal surgery (hemorrhoid banding with the 5 years of Day 1).
32. Psychosis, schizophrenia, mania, depressive disorders, history of suicide attempt or suicidal ideation, or any other psychiatric illness (with the exception of intermittent anxiety).
33. Known sensitivity to investigational product(s) or class of investigational product(s).
34. Drug or alcohol abuse within 12 months of Day 1.
35. Currently using narcotic(s) chronically.
36. Breast-feeding females.
37. Females on their menstrual cycle who cannot discern whether the bleeding is rectal bleeding or vaginal bleeding from menstruation.
38. Employees, family members, or students of the investigator or clinical site.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with cessation of bleeding by the end of Day 7 that persists for the remainder of the treatment period (through Day 14) will be analyzed as the primary endpoint | 7 days

SECONDARY OUTCOMES:
Proportion of subjects with cessation of pain by the end of Day 7 that persists for the remainder of the treatment period (through Day 14). | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Cleveland Clinic, Principal Investigator — Cleveland Clinic Weston, FL
Locations (77):
- United States (77):
  - Digestive Health, Dothan, Alabama
  - Clinical Research Associates, Huntsville, Alabama
  - Comprehensive Health Services, Phoenix, Arizona
  - Adobe, Tucson, Arizona
  - Desert Sun Clin Res, Tucson, Arizona
  - AR Gastro, Sherwood, Arkansas
  - ACRI, Anaheim, California
  - Providence Clin Res, Burbank, California
  - Med Center, Carmichael, California
  - South Orange County Surgical Group, Laguna Hills, California
  - Torrence C. R., Lomita, California
  - Premiere Clin Res, Long Beach, California
  - Facey Med Foundation, Mission Hills, California
  - Futura Research, Montebello, California
  - Community Clin Trials, Orange, California
  - Del Carmen Med Center, Reseda, California
  - MARG, San Diego, California
  - Med Center for Clinical Research, San Diego, California
  - Westlake Res, Westlake Village, California
  - Colorado Research, Salida, Colorado
  - Innovative, Clearwater, Florida
  - Avail Clin Res, DeLand, Florida
  - Eastern, Hilieah, Florida
  - Center for GI Disorders, Hollywood, Florida
  - Nature Coast Clin Res, Inverness, Florida
  - Jupiter Research, Jupiter, Florida
  - Aplusresearch, Miami, Florida
  - Kendall, Miami, Florida
  - MRA, Miami, Florida
  - Advanced Gastro Assoc, Palm Harbor, Florida
  - ICR, Sanford, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Southeast REgional Research Group, Columbus, Georgia
  - Tri County, Hartwell, Georgia
  - Southeast Regional Research Group, Savannah, Georgia
  - Pinnacle Med Inst, Overland, Kansas
  - Kentucy med Center, Lexington, Kentucky
  - Praetorian Pharmaceutical Res, Marrerro, Louisiana
  - Clinical Trials Mgmt, Metarie, Louisiana
  - Delta Research, Monroe, Louisiana
  - Women Under Study, New Orleans, Louisiana
  - Capital Digestive, Chevy Chase, Maryland
  - Meritus Center for Clin Res, Hagerstown, Maryland
  - Mid Atlantic Res Center, Hollywood, Maryland
  - Saginaw Med Res, Saginaw, Michigan
  - Gastro Assoc Western Michigan, Wyoming, Michigan
  - Gastrointestinal Associates, Jackson, Mississippi
  - Midwest Center for Clin Res, Lee's Summitt, Missouri
  - Center for Digestive & Liver Diseases, Mexico, Missouri
  - Clin Res Nevada, Las Vegas, Nevada
  - S. Jersey Gastro, Marlton, New Jersey
  - Long Island GI Group, Great Neck, New York
  - MRA NY, New York, New York
  - Ashville Gastro, Asheville, North Carolina
  - Carolinas Res Ass, Davidson, North Carolina
  - Vital, Greenboro, North Carolina
  - Carolinas Research, Harrisburg, North Carolina
  - Wake Res, Raleigh, North Carolina
  - Trial Management Associates, Wilmington, North Carolina
  - Hightop Med Res, Cincinnati, Ohio
  - Dayton Gastro, Dayton, Ohio
  - Great Lakes Gastro, Mentor, Ohio
  - Central Sooner, Norman, Oklahoma
  - Clinsearch, Chattanooga, Tennessee
  - Memphis Gastro, Germantown, Tennessee
  - Assoc of Gastro, Hermitage, Tennessee
  - Dial Research, Nashville, Tennessee
  - First Clinic, Nashville, Tennessee
  - Texas Health Research, Fort Worth, Texas
  - Amcare Research, Houston, Texas
  - Houston Gastro, Houston, Texas
  - Permian, Odessa, Texas
  - Pioneer Research, Sugarland, Texas
  - ARI, Ogden, Utah
  - ARI, Sandy City, Utah
  - New River Valley Res, Christianburg, Virginia
  - Blue Ridge Medical Center, Lyncburg, Virginia